CLINICAL TRIAL: NCT01865513
Title: POPULAR: POst-operative PULmonary Complications After Use of Muscle Relaxants in Europe - A European Prospective Multicenter Observational Study
Brief Title: POPULAR: POst-operative PULmonary Complications After Use of Muscle Relaxants in Europe
Acronym: POPULAR
Status: Completed | Type: Observational
Sponsor: European Society of Anaesthesiology (Other)
Responsible Party: Sponsor
Other Study IDs: POPULAR
Record Dates: First submitted 2013-05-28; First posted 2013-05-31 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Surgical Procedures, Operative; Anaesthesia
Keywords: Anaesthesia; Anaesthesiology; muscle Relaxants; POPULAR; postoperative pulmonary complications; Respiratory failure; Suspected pulmonary infection; Pulmonary infiltrates; Pleural effusion; Atelectasis; Pneumothorax; Bronchospasm; Aspiration pneumonitis; Cardiopulmonary oedema; European Society of Anaesthesiology; neuromuscular blockade; europe
MeSH Terms: conditions — Muscle Hypotonia; Respiratory Insufficiency; Pleural Effusion; Pulmonary Atelectasis; Pneumothorax; Bronchial Spasm; Pneumonia, Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
International multicenter observational study of a random-sample cohort of patients undergoing any in-hospital surgical procedure under general or regional anaesthesia during a continued 14-day period of recruitment.

Primary hypothesis of this study is that the use of muscle relaxants, their reversal agents, or neuromuscular monitoring increases the incidence of postoperative pulmonary complications. The secondary hypothesis is that the use of muscle relaxants increases in-hospital mortality.

DETAILED DESCRIPTION:
Overall postoperative mortality for patients undergoing non-cardiac surgery in Europe is 4% (EUSOS study). Postoperative pulmonary complications are a major factor, which increase patient morbidity and mortality (PERISCOPE study). This study is designed to evaluate the effects of management of neuromuscular blockade on postoperative pulmonary complications in a general unrestricted anaesthetized population across Europe. The investigation will be a continuation of the European EUSOS and PERISCOPE studies. Based on a well-recognised body of surrogate data, it is hypothesized that incorrect approaches to the use, monitoring, and reversal of muscle relaxants will increase the incidence of in-hospital postoperative pulmonary complications and prolong hospital stay.

The investigators will not modify a participating centre's customary management of patients. Patients with postoperative pulmonary complications will be identified by postoperative assessment and consulting medical records for events that fulfil the definition of postoperative pulmonary complications.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients undergoing any in-hospital surgical procedure under general or regional anaesthesia during the defined continued 14-day period of recruitment.

Exclusion Criteria:

1. Patients less than 18 years of age
2. Patients scheduled for local or regional anaesthesia only
3. Patient's anaesthetic procedure scheduled outside an operating room
4. Ambulatory patients = Patient planned to be discharged within 12 hours post anaesthesia
5. Patient with preoperatively intubated trachea
6. Patient from an intensive care unit (ICU)
7. Patient scheduled for additional surgical / anaesthetic procedure in the next 7 days
8. Patients who had a surgical / anaesthetic procedure within the past 7 days
9. Patient born outside the predetermined 'month(s)' allocated for the specific study centre.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Patients undergoing any in-hospital surgical procedure under general or regional anaesthesia
Sampling Method: Non-Probability Sample
Enrollment: 22000 (Actual)
Dates: Start 2014-06; Primary Completion 2015-04 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The primary study outcome parameter is the rate of post-operative pulmonary Complications (POPC). | up to 28 days after surgery
  Post-operative pulmonary Complications (POPC) is a composite of in-hospital fatal or non-fatal postoperative pulmonary events. A patient is assumed to have POPC if at least one of the following complications is documented:
  POPC is defined as a composite of in-hospital fatal or non-fatal postoperative pulmonary or respiratory events:
  Respiratory failure Suspected pulmonary infection, i.e. Suspected pulmonary infiltrates Atelectasis Aspiration pneumonitis Bronchospasm Pulmonary Oedema

SECONDARY OUTCOMES:
in-hospital mortality | up to 28 days after surgery
length of in-hospital stay | up to 28 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Blobner, M.D., Study Chair — Klinikum rechts der Isar Technische Universität München
Locations (2):
- Klinikum rechts der Isar, Technische Universität München, München, Germany
- Karolinska Institutet and Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Blobner M, Hunter JM, Meistelman C, Hoeft A, Hollmann MW, Kirmeier E, Lewald H, Ulm K. Use of a train-of-four ratio of 0.95 versus 0.9 for tracheal extubation: an exploratory analysis of POPULAR data. Br J Anaesth. 2020 Jan;124(1):63-72. doi: 10.1016/j.bja.2019.08.023. Epub 2019 Oct 10. PMID 31607388
- [Derived] Kirmeier E, Eriksson LI, Lewald H, Jonsson Fagerlund M, Hoeft A, Hollmann M, Meistelman C, Hunter JM, Ulm K, Blobner M; POPULAR Contributors. Post-anaesthesia pulmonary complications after use of muscle relaxants (POPULAR): a multicentre, prospective observational study. Lancet Respir Med. 2019 Feb;7(2):129-140. doi: 10.1016/S2213-2600(18)30294-7. Epub 2018 Sep 14. PMID 30224322